CLINICAL TRIAL: NCT04251962
Title: The Role of Epidural Opioids in Pain Management After Abdominal Surgery in Adult Patients - a Randomized Clinical Trial
Brief Title: Role of Opioids in Epidural Solutions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Israel Society of Anesthesiologists (Unknown)
Responsible Party: Principal Investigator, Barak Cohen, MD, Senior Anesthesiologist, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 0489-19-TLV
Record Dates: First submitted 2020-01-16; First posted 2020-02-05 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bupivacaine (Experimental): Epidural solution containing 0.1% bupivaacaine in normal saline
  Interventions: Drug: Bupivacaine
- Bupivacaine + Fentanyl (Experimental): Epidural solution containing 0.1% bupivacaine and 3 mcg/ml of fentanyl in normal saline
  Interventions: Drug: Bupivacaine; Drug: Fentanyl

INTERVENTIONS:
Drug: Bupivacaine — epidural solution containing bupivacaine 0.1% in normal saline
  Other Names: Marcaine
Drug: Fentanyl — Epidural solution containing fentanyl 3 mcg/ml (in addition to bupivacaine) in normal saline
  Other Names: Beatryl
  Arms: Bupivacaine + Fentanyl

SUMMARY:
It is unclear whether addition of opioids to epidural solutions for postoperative analgesia is beneficial. In this multicenter randomized double-blinded trial, we aim to test the primary hypothesis that epidural solutions containing only bupivacaine are as effective as solutions containing both bupivacaine and fentanyl in promoting analgesia in patients recovering from open abdominal surgery. We also aim to assess the incidence of epidural-induced hypotension, the difference in patient-reported opioid side-effects between the two groups. If we demonstrate no clinically important difference between the two interventions, clinicians will be able to substantially reduce the amount of opioids patients receive during their postoperative recovery, and potentially decrease the associated high incidence of opioid adverse effects in post-surgical patients.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. 18-85 years old
3. Undergoing open abdominal surgery (including colorectal, intestinal, gastric, pancreatic, hepatobiliary, urological, or gynecological surgery)
4. For which a clinical decision has been made to provide epidural analgesia preoperatively and extending to the post-operative period
5. Anticipated hospitalization of at least 2 nights

Exclusion Criteria:

1. Known allergy to bupivacaine or fentanyl
2. Chronic liver disease, defined as cirrhosis, portal hypertension, or variceal bleeding
3. Patients under chronic alpha-blocking agents for hypertension
4. Clinical contraindications to epidural introduction, as judged by the anesthesia provider (thrombocytopenia, un-interrupted anticoagulation, clinically-significant atrio-ventricular conduction block, etc.)
5. Pregnant women

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2022-03-02 (Actual)

PRIMARY OUTCOMES:
Postoperative analgesia | 48 postoperative hours
  A joint outcome of the difference in average pain score and a ratio of opioid consumption (in mg morphine equivalents) between the 2 study groups

SECONDARY OUTCOMES:
Clinically significant postoperative hypotension | 48 postoperative hours
  Number of participants experiencing a composite of use of IV fluid boluses prescribed for hemodynamic support; sympathomimetic drugs administration; and holding or early discontinuation of the epidural infusion in order to recover blood pressure.

OTHER OUTCOMES:
Recovery of gastrointestinal function | Throughout the postoperative hospital stay, up to 30 days
  Time to first postoperative bowel movement
Opioid-related side effects | 48 postoperative hours
  A composite of opioid-related side-effects as measured by the Opioid-Related Symptom Distress Scale (OR-SDS) questionnaire (higher scores represent more side-effects and related distress, scores are given on multiple dimensions)

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Anesthesia, Pain and Critical Care, Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No